CLINICAL TRIAL: NCT01609101
Title: Oropharyngeal Space in Videolaryngoscopy: a Randomised Crossover Trial Measuring Remaining Space Adjacent to the Videolaryngoscope Blade
Brief Title: Oropharyngeal Space in Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Barbe Pieters, Principal Investigator, Catharina Ziekenhuis Eindhoven
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: M12-1210; M12-1210 (Other: Catharina Ziekenhuis Eindhoven)
Record Dates: First submitted 2012-05-24; First posted 2012-05-31 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Abrasion of Soft Palate; Intubation Complication
Keywords: Videolaryngoscopy; Palatopharyngeal distance; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Coopdech® videolaryngoscope (Other)
  Interventions: Device: Coopdech® videolaryngoscope
- C-MAC® videolaryngoscope (Other)
  Interventions: Device: C-MAC ® videolaryngoscope
- McGrath® Series 5 videolaryngoscope (Other)
  Interventions: Device: McGrath® Series 5 videolaryngoscope
- Glidescope® Cobalt videolaryngoscope (Other)
  Interventions: Device: Glidescope® Cobalt videolaryngoscope
- King Vision® videolaryngoscope (Other)
  Interventions: Device: King Vision® videolaryngoscope
- Venner® videolaryngoscope (Other)
  Interventions: Device: Venner® videolaryngoscope
- McGrath MAC® videolaryngoscope (Other)
  Interventions: Device: McGrath® MAC

INTERVENTIONS:
Device: C-MAC ® videolaryngoscope — C-MAC ® videolaryngoscope
  Other Names: C-MAC ® videolaryngoscope (Karl Storz, Tuttlingen, Germany)
  Arms: C-MAC® videolaryngoscope
Device: Coopdech® videolaryngoscope — Coopdech® videolaryngoscope
  Other Names: Coopdech® videolaryngoscope (Daiken Medical, Osaka, Japan)
  Arms: Coopdech® videolaryngoscope
Device: McGrath® Series 5 videolaryngoscope — McGrath® Series 5 videolaryngoscope
  Other Names: McGrath® Series 5 (Aircraft Medical, Edinburgh, UK)
  Arms: McGrath® Series 5 videolaryngoscope
Device: Glidescope® Cobalt videolaryngoscope — Glidescope® Cobalt videolaryngoscope
  Other Names: Glidescope® Cobalt (Verathon, Bothell, USA)
  Arms: Glidescope® Cobalt videolaryngoscope
Device: King Vision® videolaryngoscope — King Vision® videolaryngoscope
  Other Names: King Vision® videolaryngoscope (King Systems, Noblesville, IN, USA)
  Arms: King Vision® videolaryngoscope
Device: Venner® videolaryngoscope — Venner® videolaryngoscope
  Other Names: Venner® videolaryngoscope (Venner Medical, Singapore, Republic of Singapore)
  Arms: Venner® videolaryngoscope
Device: McGrath® MAC — McGrath® MAC (Aircraft Medical, Edinburgh, UK)
  Other Names: McGrath® MAC (Aircraft Medical, Edinburgh, UK)
  Arms: McGrath MAC® videolaryngoscope

SUMMARY:
In this randomised crossover trial we measure the space between the right side of the laryngoscope blade and the right palatopharyngeal wall in a cohort of ASA I-III patients with a normal mouth opening. We compare the remaining spaces for seven different videolaryngoscopes and compare these to a classic Macintosh laryngoscope.

DETAILED DESCRIPTION:
Intubation using indirect videolaryngoscopy has many advantages over classic direct laryngoscopy using the Macintosh laryngoscope. There are many different videolaryngoscopes available, and the blade differs largely between videolaryngoscopes. Different size and angles of blades may have an impact on the space available for insertion of the endotracheal tube. The space between the blade and the palatopharyngeal wall may be reduced significantly, so that there is less room in the mouth to insert an endotracheal tube. Positioning and manoeuvring of the endotracheal tube may consequently be more difficult and may traumatize the pharynx as was described in a few case reports, especially when an endotracheal tube with a rigid stylet inserted was used.

ELIGIBILITY:
Inclusion Criteria:

* Informed patient consent
* ASA I - III
* Age > 18 years
* Elective surgery, other than head and/or neck surgery
* Pre-operative Mallampati I - III
* BMI < 35 kg/m2
* Fasted (≥6 hours)

Exclusion Criteria:

* No informed patient consent
* ASA ≥ IV
* Age < 18 year
* Emergency surgery, surgery of head and/of neck
* Locoregional anaesthesia
* Pre-operative Mallampati IV
* BMI > 35 kg/m2
* Fasted < 6 hours
* Pre-operative expected difficult airway (restrict neck movement, thyromental distance < 65mm, retrognathia)
* Bad, fragile dentition
* Dental crowns and/or fixed partial denture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Palatopharyngeal distance | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Two laryngoscopes (one classic direct laryngoscope and one indirect videolaryngoscope) will subsequently be inserted into the patient's mouth at random order. With each laryngoscope the horizontal distance between the laryngoscope blade and mid-palatopharyngeal fold will be measured using an mm ruler.

SECONDARY OUTCOMES:
Difference in palatopharyngeal distance between videolaryngoscope and classic Macintosh laryngoscope | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Investigating how this space differs from the space that remains on the right side of the blade of the classic Macintosh laryngoscope and the palatopharyngeal wall in the same cohort of patients.
Difference in palatopharyngeal distance between videolaryngoscopes | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Comparing the difference in remaining palatopharyngeal space between the different videolaryngoscopes.
Cormack-Lehane score | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Registering difficulty of intubation (Cormack-Lehane score)
Successful intubation | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Registering the number of successful intubations.
Use of rigid stylet | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Use of rigid stylet during intubation
Number of attempts | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Number of intubation attempts
Time until picking up endotracheal tube | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Time until picking up endotracheal tube
Epiglottic down-folding | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Occurrence of epiglottic down-folding
Complications | Participants will be followed during induction of anesthesia, an expected average of 10 min
  Any complication that occurs during intubation will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Andre A van Zundert, MD PhD FRCA, Study Director — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] Cooper RM. Complications associated with the use of the GlideScope videolaryngoscope. Can J Anaesth. 2007 Jan;54(1):54-7. doi: 10.1007/BF03021900. PMID 17197469
- [Background] Cross P, Cytryn J, Cheng KK. Perforation of the soft palate using the GlideScope videolaryngoscope. Can J Anaesth. 2007 Jul;54(7):588-9. doi: 10.1007/BF03022329. No abstract available. PMID 17602049
- [Background] Hirabayashi Y. Pharyngeal injury related to GlideScope videolaryngoscope. Otolaryngol Head Neck Surg. 2007 Jul;137(1):175-6. doi: 10.1016/j.otohns.2007.02.038. No abstract available. PMID 17599592
- [Background] Manickam BP, Adhikary SD. Re: Soft palate perforation during orotracheal intubation facilitated by the GlideScope videolaryngoscope. J Clin Anesth. 2008 Aug;20(5):401-402. doi: 10.1016/j.jclinane.2008.01.009. No abstract available. PMID 18761255
- [Background] Vincent RD Jr, Wimberly MP, Brockwell RC, Magnuson JS. Soft palate perforation during orotracheal intubation facilitated by the GlideScope videolaryngoscope. J Clin Anesth. 2007 Dec;19(8):619-21. doi: 10.1016/j.jclinane.2007.03.010. PMID 18083477